CLINICAL TRIAL: NCT02188290
Title: An Observational Cohort Study on Transplant-Related Mortality in Patients Receiving Either a Hematopoietic Stem Cell Transplantation Without ATIR or an Umbilical Cord Blood Transplantation
Brief Title: Transplant-Related Mortality in Patients Undergoing a Peripheral Blood Stem Cell Transplantation or an Umbilical Cord Blood Transplantation
Status: Completed | Type: Observational
Sponsor: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-AIR-006
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: Haploidentical donor; Unrelated donor; Umbilical cord blood; Graft versus host disease; Transplant-related mortality; Hematologic malignancy; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- HAPLO group: Control group of all eligible patients who received an HSCT from a haploidentical donor without ATIR administration between 1 January 2006 and 30 June 2013
- MUD group: Control group of eligible patients who received an HSCT from a fully matched unrelated donor between 1 January 2010 and 31 December 2012
- MMUD group: Control group of eligible patients who received an HSCT from a 1-locus mismatched unrelated donor between 1 January 2010 and 31 December 2012
- UCB group: Control group of eligible patients who received a double umbilical cord blood transplantation between 1 January 2010 and 31 December 2012

SUMMARY:
Study CR-AIR-006 is a part of the ATIR clinical development plan and will provide control data for patients treated with ATIR in clinical studies (e.g. study CR-AIR-007).

ELIGIBILITY:
Inclusion Criteria:

* Any of the following hematologic malignancies:

  * Acute myeloid leukemia (AML) in remission at the time of the transplantation
  * Acute lymphoblastic leukemia (ALL) in remission at the time of the transplantation
  * Myelodysplastic syndrome (MDS)
* Patient received any of the following transplantations:

  * Allogeneic T-cell depleted HSCT without ATIR administration from a haploidentical donor between 1 January 2006 and 30 June 2013 (HAPLO group)
  * Allogeneic HSCT from a fully matched or 1-locus mismatched unrelated donor between 1 January 2010 and 31 December 2012 (MUD/MMUD groups)
  * Double umbilical cord blood transplantation between 1 January 2010 and 31 December 2012 with no more than 2 human leukocyte antigen (HLA)-mismatches at HLA-A, B, and/or -DR between each of the units and the recipient (UCB group)
* Male or female, age ≥ 18, ≤ 65 years.

Exclusion Criteria:

* Allogeneic stem cell transplantation prior to the transplantation qualifying for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having received a haploidentical hematopoietic stem cell transplantation (HSCT) between 1 January 2006 and 30 June 2014, an HSCT from an unrelated donor between 1 January 2010 and 31 December 2012, or a double UCB transplantation between 1 January 2010 and 31 December 2012 will be selected from the centers that enrolled patients in study CR-AIR-004 and/or study CR-AIR-007.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Transplant-related mortality | Up to 12 months after the transplantation

SECONDARY OUTCOMES:
Overall survival | Up to 12 months after the transplantation
Incidence of acute and chronic graft versus host disease | Up to 12 months after the transplantation
Progression-free survival | Up to 12 months after the transplantation
Severity of acute and chronic graft versus host disease | Up to 12 months after the transplantation
Relapse-related mortality | Up to 12 months after the transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Rovers, MD, Study Chair — Kiadis Pharma
Locations (9):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States
- Belgium (3):
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gasthuisberg, Leuven
- Canada (2):
  - Hamilton Niagara Regional Haemophilia Centre, Hamilton, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- Universitätsklinikum Würzburg, Würzburg, Germany
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Hammersmith Hospital, London, United Kingdom